CLINICAL TRIAL: NCT05586750
Title: Clinical Trial to Determine the Effects of Statins on Brain Health - STAREE-Mind Imaging Substudy
Brief Title: Statins in Reducing Events in the Elderly Mind (STAREE-Mind) Imaging Substudy
Acronym: STAREE-Mind
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Monash University (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Principal Investigator, Joanne Ryan, Professor, Monash University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2006611
Record Dates: First submitted 2022-10-10; First posted 2022-10-19 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2024-11

CONDITIONS: Dementia, Mixed; Dementia, Vascular; Dementia of Alzheimer Type; Cognitive Decline; White Matter Hyperintensity; Aging; Neuro-Degenerative Disease
Keywords: White matter mean diffusivity; Perivascular space; Free water; White matter hyperintensity
MeSH Terms: conditions — Mixed Dementias; Dementia, Vascular; Cognitive Dysfunction | interventions — Atorvastatin; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- STAREE Statin group (Experimental)
  Interventions: Drug: Atorvastatin 40 Mg Oral Tablet
- STAREE Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin 40 Mg Oral Tablet — 40 mg atorvastatin (2 x 20 mg atorvastatin daily), taken orally
  Arms: STAREE Statin group
Drug: Placebo — 2 x 20mg placebo (daily), taken orally. Identical appearance to study drug
  Arms: STAREE Placebo group

SUMMARY:
The STAREE-Mind imaging sub-study will examine the effect of statin treatment over a 4-year period, compared with placebo, on markers of brain health.

DETAILED DESCRIPTION:
STAREE-Mind imaging is a sub-study nested in the Statins in Reducing Events in the Elderly (STAREE) double blind randomised placebo-controlled trial. STAREE is investigating whether statins can prolong good health and maintain independence amongst older people and is enrolling. STAREE-Mind imaging aims to recruit a sub-group of 340 participants, and will involve an additional suite of brain imaging in these participants, at recruitment (before medication is commenced) and at 4 years follow-up. It will provide crucial information about the clinical effects of statins on brain health in older individuals.

ELIGIBILITY:
Inclusion Criteria:

* Participants in the STAREE RCT and eligible for randomisation to study medication.
* Men and women
* Aged ≥70 years
* Living independently in the community
* Willing and able to provide informed consent and agree to participate in brain neuroimaging.
* Able to attend one of the 2 sites (in Melbourne and Brisbane) where the imaging will take place.

Exclusion Criteria:

* Contraindications to have magnetic resonance neuroimaging performed.
* History of invasive brain surgery or known structural bran abnormalities.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 341 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Free water | Change from baseline to four years
  Multi-compartment free water quantitation from brain diffusion-weighted MRI
White matter hyperintensity volume | Change from baseline to four years
  From brain FLAIR MRI

OTHER OUTCOMES:
Cortical thickness | Change from baseline to four years
  Cortical thickness as measured by T1-weighted structural MRI.
Hippocampal volume | Change from baseline to four years
Microbleeds and lacunae | Change from baseline to four years
Prefrontal cortex cerebral perfusion | Change from baseline to four years
  Prefrontal cortex cerebral perfusion as measured by pseudo-continuous arterial spin labelling (pCASL) MRI.
Whole-brain white matter fractional anisotropy | Change from baseline to four years
  Whole-brain white matter fractional anisotropy as measured by diffusion-weighted imaging (DWI) MRI.
Peri-vascular space volume | Change from baseline to four years
  From brain T1-weighted MRI

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Zoungas, MBBS, FRACP, Principal Investigator — Monash University
Locations (2):
- Australia (2):
  - Herston Imaging Research Facility (HIRF), Herston, Queensland
  - Monash Biomedical Imaging (MBI), Clayton, Victoria

IPD SHARING:
Plan to Share IPD: Yes
After publication of the trial outcomes, the de-identified data will be available to approved researchers through a secure portal.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Harding IH, Ryan J, Heritier S, Spark S, Flanagan Z, McIntyre R, Anderson CS, Naismith SL, Chong TT, O'Sullivan M, Egan G, Law M, Zoungas S. STAREE-Mind Imaging Study: a randomised placebo-controlled trial of atorvastatin for prevention of cerebrovascular decline and neurodegeneration in older individuals. BMJ Neurol Open. 2023 Oct 31;5(2):e000541. doi: 10.1136/bmjno-2023-000541. eCollection 2023. PMID 37920607